CLINICAL TRIAL: NCT00316849
Title: A Phase I Study of CCI-779, and Temozolomide in Combination With Radiation Therapy in Glioblastoma Multiforme
Brief Title: Temsirolimus, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00642; N027D; CDR0000467232; NCCTG-N027D; U10CA025224 (NIH)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Chemotherapy, Adjuvant; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; temsirolimus; Sirolimus; Temozolomide

ARMS (1):
- Treatment (temsirolimus, temozolomide, radiation therapy) (Experimental): GROUP 1: (temsirolimus with radiation and temozolomide) Patients receive temsirolimus IV over 30 minutes once weekly. Beginning 7-10 days later, patients also receive oral temozolomide daily and undergo concurrent 3-D conformal radiotherapy or intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks. Patients with stable or responding disease proceed to adjuvant therapy. GROUP 2: (radiation and temozolomide) Patients receive oral temozolomide daily and undergo concurrent 3-D conformal radiotherapy or intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks. Patients with stable or responding disease proceed to adjuvant therapy. ADJUVANT THERAPY: Beginning 4-6 weeks after the completion of chemoradiotherapy patients receive oral temozolomide on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: pharmacological study; Procedure: adjuvant therapy; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy; Drug: temsirolimus; Drug: temozolomide

INTERVENTIONS:
Other: pharmacological study
  Other Names: pharmacological studies
Procedure: adjuvant therapy
Radiation: 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Radiation: intensity-modulated radiation therapy
  Other Names: IMRT
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Drug: temozolomide — Given orally
  Other Names: SCH 52365; Temodal; Temodar; TMZ

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus when given together with temozolomide and radiation therapy in treating patients with newly diagnosed glioblastoma multiforme. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving temsirolimus together with temozolomide and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of temsirolimus when administered with temozolomide in combination with radiotherapy followed by adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme.

II. Assess and describe the adverse events associated with this regimen in these patients.

III. Evaluate the early response to therapy in these patients using an automated morphological MRI change detector and physiological MRI techniques, including diffusion-weighted imaging, perfusion-weighted imaging, and chemical shift imaging.

SECONDARY OBJECTIVES:

I. Determine the inhibition status of mTOR signaling pathways in peripheral blood mononuclear cells in patients treated with this regimen.

II. Identify potential pharmacokinetic interactions between temozolomide and temsirolimus.

III. Correlate, preliminarily, survival, progression-free survival, and response with pre-treatment tumor tissue molecular markers in these patients.

OUTLINE: This is a multicenter, dose-escalation study of temsirolimus. Patients are assigned to 1 of 2 treatment groups.

GROUP 1: (temsirolimus with radiation and temozolomide) Patients receive temsirolimus IV over 30 minutes once weekly. Beginning 7-10 days later, patients also receive oral temozolomide daily and undergo concurrent 3-D conformal radiotherapy or intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks. Patients are evaluated 4-6 weeks after completion of chemoradiotherapy. Patients with stable or responding disease proceed to adjuvant therapy. Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience a dose-limiting toxicity. At least 6 patients are treated at the MTD.

GROUP 2: (radiation and temozolomide) Patients receive oral temozolomide daily and undergo concurrent 3-D conformal radiotherapy or intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks. Patients are evaluated 4-6 weeks after completion of chemoradiotherapy. Patients with stable or responding disease proceed to adjuvant therapy.

ADJUVANT THERAPY: Beginning 4-6 weeks after the completion of chemoradiotherapy patients receive oral temozolomide on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo blood collection for immune monitoring and translational/pharmacologic studies. After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme (GBM)

  * Gliosarcoma and other grade 4 astrocytoma variants (e.g., giant cell glioblastoma) allowed
* Newly diagnosed disease

  * Has undergone surgical resection or biopsy of the tumor at least 1 week but no more than 6 weeks ago
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2.5 times upper limit of normal (ULN)
* Cholesterol < 350 mg/dL
* Triglycerides < 400 mg/dL
* AST ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergy or intolerance to dacarbazine
* No ongoing or active infection
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No gastrointestinal tract disease affecting ability to take oral medication or requiring IV alimentation
* No significant traumatic injury within the past 21 days
* No active, uncontrolled peptic ulcer disease
* No other active cancers requiring therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Willing and able to comply with antibiotic prophylaxis with either trimethoprim/sulfamethoxazole (daily or 3 times per week) or monthly IV pentamidine combined with daily levofloxacin
* No prior chemotherapy for any brain tumor
* No prior temozolomide or mTOR inhibitor therapies
* No prior cranial radiotherapy
* More than 21 days since prior major surgery (excluding neurosurgical biopsy or resection of GBM)
* No prior surgical procedures affecting absorption
* No concurrent enzyme-inducing anticonvulsants, including any of the following:

  * Carbamazepine
  * Phenytoin
  * Phenobarbital
  * Primidone
* No other concurrent investigational agents
* Not receiving warfarin prior to study registration

  * Concurrent warfarin allowed if patients develop an indication for it while enrolled on the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-05; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD), determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | Up to 24 weeks
Time to treatment related toxicity as assessed by hematologic measures and CTCAE v3.0 | From registration to documentation of toxicity, up to 5 years
Time to treatment related toxicity greater than grade 3, assessed by CTCAE v3.0 | From registration to documentation of toxicity, up to 5 years
Time to progression | From registration to documentation of progression, up to 5 years
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by patient, up to 5 years
  Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals.The effect of dose and ancillary dichotomized covariates such as gender or age (<50 years versus 50+ years) will be explored using logrank testing involving one covariate at a time.
Response to therapy associated with patient outcome, as assessed by automated morphological MRI change detector and physiological MRI techniques, including diffusion-weighted imaging, perfusion-weighted imaging, and chemical shift imaging | Up to 5 years
  Logistic regression and Cox proportional hazards models will be used to determine the association between changes in tumor volume (as assessed by a software package) and tumor response and 12-month survival (logistic regression) and progression-free and overall survival (Cox proportional hazards models).

CONTACTS AND LOCATIONS:
Overall Officials: Jann Sarkaria, Principal Investigator — North Central Cancer Treatment Group
Locations (11):
- United States (11):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Altru Cancer Center, Grand Forks, North Dakota